CLINICAL TRIAL: NCT01009619
Title: Randomized Double-blind Placebo-controlled Prevention Trial of Azithromycin in Lung Transplantation.
Brief Title: Azithromycin in Bronchiolitis Obliterans Syndrome
Acronym: AZI001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University Hospital, Gasthuisberg (Other); Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Prof. Dr. GM. Verleden, KULeuven and University Hospital Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZI001; EudraCT ref. 2005-003893-46 (Registry Identifier: ISRCTN36220396)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Bronchiolitis Obliterans Syndrome; Graft Rejection; Lymphocytic Bronchiolitis; Respiratory Infection
Keywords: Bronchiolitis Obliterans Syndrome; Acute allograft Rejection; Lymphocytic bronchiolitis; Respiratory infection; Survival; Mortality; Pulmonary function; FEV1; Broncho-alveolar lavage; Neutrophils; Interleukin; Culture; Azithromycin
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Respiratory Tract Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (Experimental): 250 mg daily for 5 days, followed by 250 mg three times a week (Mon.-Wed.-Fri.) until the end of study
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): PLacebo daily for 5 days, followed by placebo three times a week (Mon.-Wed.-Fri.) until end of study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 250 mg daily during 5 days followed by 250 mg three times a week on Mon., Wed. and Fri. during study-period.
  Other Names: Zitromax (Azithromycin Dihydrate, Pfizer, ZTM250)
  Arms: Azithromycin
Drug: Placebo — Placebo once daily during 5 days, followed by one placebo three times a week on Mon., Wed. and Fri during rest of study-period.
  Other Names: Lactose monohydricum Ph.Eur. (Fagron)
  Arms: Placebo

SUMMARY:
Preventive treatment with azithromycin reduces the prevalence fo Bronchiolitis Obliterans Syndrome after lung transplantation.

DETAILED DESCRIPTION:
* Prospective, interventional, randomized, double-blind, placebo-controlled trial.
* Clinical setting (tertiary University Hospital).
* Investigator-driven, no pharmaceutical sponsor.
* Lung transplant recipients.
* Add-on of study-drug (placebo or azithromycin) to 'standard of care' (standardized, routine immunosuppressive and infectious prophylactic protocol).
* 1:1 inclusion ratio (placebo:azithromycin).
* Randomisation at discharge after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Stable LTx recipients at discharge after transplantation.
* Signed informed consent
* Adult (age at least 18 years old at moment of transplantation)
* Able to take oral medication

Exclusion Criteria:

* Prolonged and/or complicated ICU-course after transplantation.
* Early (<30 days post-transplant) post-operative death
* Major suture problems (airway stenosis or stent)
* Retransplantation (lung)
* Previous transplantation (solid organ)
* Multi-organ transplantation (lung+ other solid organ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geert M Verleden, Prof. Dr., Principal Investigator — KULeuven and University Hospitals Leuven
Locations (1):
- Katholieke Universiteit Leuven and University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Derived] Ruttens D, Verleden SE, Vandermeulen E, Bellon H, Vanaudenaerde BM, Somers J, Schoonis A, Schaevers V, Van Raemdonck DE, Neyrinck A, Dupont LJ, Yserbyt J, Verleden GM, Vos R. Prophylactic Azithromycin Therapy After Lung Transplantation: Post hoc Analysis of a Randomized Controlled Trial. Am J Transplant. 2016 Jan;16(1):254-61. doi: 10.1111/ajt.13417. Epub 2015 Aug 4. PMID 26372728
- [Derived] Vos R, Vanaudenaerde BM, Verleden SE, De Vleeschauwer SI, Willems-Widyastuti A, Van Raemdonck DE, Schoonis A, Nawrot TS, Dupont LJ, Verleden GM. A randomised controlled trial of azithromycin to prevent chronic rejection after lung transplantation. Eur Respir J. 2011 Jan;37(1):164-72. doi: 10.1183/09031936.00068310. Epub 2010 Jun 18. PMID 20562124

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 40 | 43
Completed | 40 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 42 | 80
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 51.2 (0) | 50.9 (0) | 51.1 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  Belgium | 40 | 43 | 83

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Bronchiolitis Obliterans Syndrome (BOS)
Description: BOS was defined as a sustained decrease in forced Expiratory Volume in one second (FEV1) of at least 20% from the patient's maximum post-operative values in the absence of other causes.
Time Frame: 2 years post-transplant
Population: intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
participants | 5 [0 to 0] | 19 [0 to 0]

2. Primary Outcome: Overall Survival
Description: Survival data were obtained using all-cause mortality information in the Leuven University Hospital transplant database, in which all our lung transplant recipients since 1991 are registered. For the end-point of all-cause mortality, survival times were not censored at retransplantation or at study-discontinuation if these preceded death, or else at 2 years after transplantation.
Time Frame: 2 years post-transplant
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
participants | 6 | 8

3. Secondary Outcome: Acute Rejection Incidence Rate
Description: Bronchoscopy and broncho-alveolar lavage (BAL) was routinely performed at discharge, 3, 6, 12, 18, 24 months post-transplantation and later at intervals of 1 year, or in case of clinically suspected acute allograft rejection, infection or chronic rejection. Transbronchial biopsies were routinely performed at discharge and 3 months post-transplant or in case of suspected acute rejection, infection or chronic rejection. Biopsies were graded according to the 1996 ISHLT-guidelines (grade A0-4 with concomitant B0-4), as well as assessed for other interstitial lesions of the pulmonary graft.
Time Frame: 2 years post-transplant
Measure: Mean (Standard Deviation); unit: incidence rate (events/person per year)
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
incidence rate (events/person per year) | 0.86 (1.53) | 0.78 (1.17)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; The frequency or rate of specific events (i.e. acute rejection, cytomegalovirus (CMV) and non-CMV infections) was calculated by determining the number of events per year of study time for each subject, correcting for CMV-mismatch status; Test type: Superiority or Other; p < 0.05, Chi-squared, Corrected

4. Secondary Outcome: Infection Incidence Rate
Description: Cytomegalovirus (CMV)-status was assessed on on every broncho-alevolar lavage sample and by serum CMV DNA at weekly intervals during hospitalization and thereafter at each outpatient evaluation or hospital admission. Immunohistochemical staining for CMV was performed on transbronchial biopsies in case of clinical suspicion of infection (i.e. dyspnea, cough, sputum, fever, increased plasma C-reactive protein, new chest radiograph infiltrates, or a decrease of at least 10% in peak expiratory flow (PEF) as measured by patient's peak flow measurements.
Time Frame: 2 years post-transplant
Population: intention to treat
Measure: Mean (Standard Deviation); unit: incidence rate (events/person per year)
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
incidence rate (events/person per year) | 0.95 (1.4) | 0.73 (1.42)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.05, Chi-squared, Corrected

5. Secondary Outcome: Pulmonary Function
Description: Spirometry (Masterscreen, Jaeger, Hoechberg, Germany) was performed at twice weekly intervals for the first 2 postoperative months, thereafter at weekly to biweekly intervals until 6 months post-transplantation, then every 2 to 4 weeks until the first postoperative year and afterwards life-long at intervals of 2 to 3 months according to American Thoracic Society standards and forced expiratory volume in one second (FEV1) expressed in terms of the percentage of predicted values.
Time Frame: during first two years post-transplant
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
percent predicted | 81.11 (20.31) | 75.28 (25.31)

6. Secondary Outcome: Broncho-alveolar (BAL) Neutrophilia
Description: BAL was performed with two 50 mL aliquots of sterile saline at room temperature. Five mL of the recovered BAL fluid was sent for microbiological and virological assessment, whereas the remaining fluid was analysed for cell counts after a cytospin was made in a Shandon cytocentrifuge and stained with May-Grünwald-Giemsa. Differential cell counts were determined by counting at least 300 cells.
Time Frame: during first two years post-transplant
Measure: Mean (Standard Deviation); unit: percent cells
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
percent cells | 9.68 (18.20) | 15.73 (25.36)

7. Secondary Outcome: Plasma C-reactive Protein (CRP) Levels
Description: Plasma C-reactive protein (CRP) levels were assessed using Tina-quant CRP latex assay, Roche, Mannheim, Germany; sensitivity threshold of 1 mg/L, upper limit of normal 5 mg/L.
Time Frame: during the first two years post-transplant
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 40 | 43
mg/L | 7.06 (16.97) | 10.02 (17.51)

ADVERSE EVENTS:
Time Frame: A study-nurse verified compliance and possible adverse events at each contact with patients during routine follow-up visits at the outpatient clinic or hospital-admissions during the first two years post-transplant.
Description: Definition for adverse events:
  Serious adverse events: allergic (rash, urticaria, Stevens-Johnson syndrome, angioneurotic edema or anaphylaxis), cardiac (ventricular tachycardia or Torsades de Pointes), neurologic (convulsions).
  Other adverse events: gastro-intestinal (nausea, dyspepsia, pain or cramps, diarrhea or pseudomembranous colitis).
Arm/Group | Azithromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 3/40 | 0/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=40) | Placebo (N=43)
nausea and diarrhea after intake of study drug (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes